CLINICAL TRIAL: NCT02932813
Title: The Effects of a Translational Health After School Program on Health-Related Knowledge/Behaviors and Exercise Perception in Minority Children
Brief Title: Translational Health After School Program on Health-Related Knowledge/Behaviors and Exercise Perception
Acronym: THINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Sherman Fairchild Foundation (Unknown)
Responsible Party: Principal Investigator, Arlette Perry, Professor of Kinesiology and Sport Sciences, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20160719
Record Dates: First submitted 2016-09-01; First posted 2016-10-13 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Changes in Physical Fitness; Changes in Diet, Food, and Nutrition Habits; Changes in Child Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): THINK intervention:
  The program will have activity and fitness sessions lasting two hours, three times a week for a total of nine months. Sessions will include theory, clinical laboratory activities, and physically active games to facilitate a fun environment to enhance physical and health-related fitness, improve nutrition and exercise knowledge and behaviors, and exercise enjoyment and self-confidence.
  Interventions: Behavioral: THINK Program
- Control Group (No Intervention): This group will receive the traditional YMCA SPARK after-school program. They will undergo the same pre, mid, and post testing protocol as the intervention group, but will not receive the THINK program.

INTERVENTIONS:
Behavioral: THINK Program — Lessons and laboratory sessions will be 60 minutes, followed by physical activity sessions lasting 60 minutes. Laboratory activities include assessing heart rate, making healthy meals, learning portion sizes, brain challenges, and more. To improve physical activity participation, a wide selection of developmentally appropriate and multiculturally sensitive activities will be offered, such as sports, games, obstacle courses, and dance.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to examine the effects of a translational health in nutrition and kinesiology (THINK) after school program on physical variables, nutrition and exercise knowledge base/behaviors, and exercise enjoyment and confidence.

Partnering with the YMCA investigators in the Kinesiology and Sport Sciences department at the University of Miami will set up the after-school THINK program offered three afternoons per week for nine months in two experimental and two control schools. The schools will consist of minority elementary school students (predominantly Hispanic and Black) in the South Florida area. The control schools will receive baseline, mid-year and follow-up testing nine months later, but will not go through the THINK program. They will instead go through their standard YMCA after school Sports, Play, and Active Recreation for Kids (SPARK) program.

DETAILED DESCRIPTION:
Two- thirds of American adults are overweight or obese, and that number continues to rise. Thus, it is not surprising that the prevalence of overweight/obesity has more than doubled in school children and tripled in adolescents. Concomitant with the rise in obesity has been a significant decrease in physical fitness levels (1,2). At least one study has shown the youth of today demonstrate lower aerobic fitness levels than their parents (3). Low aerobic fitness levels are most prevalent among Hispanic and Black (non-Hispanic) minority youth. No doubt the increases in TV viewing, computer time and technology have contributed to the increase in sedentary habits and decline in physical activity levels (4).

The THINK program translates fitness and health-related information into knowledge and skills that children can understand and incorporate into their own personal health and lifestyle behaviors. The program is unique in that it combines educational and hands-on clinical experiences with physical activity and exercise. The goal is to promote healthier, more active children of today who demonstrate improved levels of physical fitness, exercise knowledge, and enjoyment of tomorrow.

Each unit in the THINK program has three components: a seminar on the scientific aspects of a health-related theme, clinical experiences related to the theme, and related physical activities performed in the field. The THINK seminars engage students by getting them up and moving, while asking questions that prompt them to think creatively to come up with their own answers. Clinical experiences reinforce the educational themes allowing children to learn more about their bodies, how it functions, and how it adapts through various movement exercises. Finally, games and enjoyable physical activities round out the program contributing to enhanced motor skill development and improved physical fitness levels.

The THINK program will begin with a series of baseline physical assessments comprising both heath and performance-related physical fitness. Participants will also receive a quiz on nutrition and exercise-related information and two surveys regarding nutritional behaviors and physical activity levels. They will be asked to complete one survey on exercise enjoyment and self-confidence. Parents will also be asked to complete a survey each on their child's nutritional habits. This will be done in two experimental and two control YMCA after school programs comprising primarily minority (Hispanic and Black) participants. Testing will again take place midway through the program and at the conclusion of the program nine months later. The control group will not go through the THINK program but will instead go through the traditional SPARK curriculum.

The purpose of the study is to determine whether the THINK program results in improvements in physical fitness, nutrition and exercise knowledge/habits, and exercise enjoyment and self-confidence above that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Children in grades 3-5 (aged 8-12)
* enrolled in a YMCA after-school program

Exclusion Criteria:

* Inability to perform physical activity
* Any cardiovascular, metabolic, or neurological disorders that would affect the child's ability to participate in the program or in testing.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Resting Measures | Baseline, at 4 months, and at 9 months
  Resting heart rate and blood pressure will be assessed using an automatic blood pressure cuff.
Aerobic fitness | Baseline, at 4 months, and at 9 months
  An NIH 2 minute walk test will be used to assess aerobic fitness.
Agility and speed | Baseline, at 4 months, and at 9 months
  A shuttle run will be used to assess agility and speed.
Upper-body strength and endurance | Baseline, at 4 months, and at 9 months
  A hand-grip dynamometer will be used to assess upper body strength and endurance
Abdominal strength and endurance | Baseline, at 4 months, and at 9 months
  A one minute curl-up (sit up) will be used to assess abdominal strength and endurance.
Lower body power | Baseline, at 4 months, and at 9 months
  The height of a vertical jump test will be used to assess lower body power.
Flexibility | Baseline, at 4 months, and at 9 months
  A lower body sit and reach test will be used to assess flexibility.

SECONDARY OUTCOMES:
Body Composition | Baseline, at 4 months, and at 9 months
  Electrical impedance and 3 site Skinfolds
Body fat distribution | Baseline, at 4 months, and at 9 months
  Waist and hip circumference will be measured
Exercise Enjoyment and Confidence | Baseline, at 4 months, and at 9 months
  A modified Exercise Enjoyment Scale and a modified Exercise Self-Confidence Scale will be given
Knowledge/Behaviors/Habits | Baseline, at 4 months, and at 9 months
  International Physical Activity Questionnaire (IPAQ) and The CATCH Kids Club questionnaire will be given.
Nutritional survey | Baseline, at 4 months, and at 9 months
  A parental survey of family nutrition behaviors will be given and An Exercise Physiology and Nutrition Knowledge Base Test

CONTACTS AND LOCATIONS:
Overall Officials: Arlette Perry, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes